CLINICAL TRIAL: NCT01795157
Title: Computer Based Assessment and Treatment
Acronym: COMBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/859
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Neoplasms; Pain
Keywords: decision support systems, clinical; decision making, computer assisted; evidence based practice; practice guidelines as topic
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCADSS (Experimental): questionnaire completed using i-Pad
  Interventions: Device: CCADSS
- pen-paper (Active Comparator): Questionnaire completed using pen and paper
  Interventions: Device: pen-paper

INTERVENTIONS:
Device: CCADSS — Questionnaire is transferred wireless to the physician's PC
  Arms: CCADSS
Device: pen-paper — Questionnaire completed and transferred to the physician using standard methods
  Arms: pen-paper

SUMMARY:
This study aims to investigate computer based symptom assessment in an outpatient cancer population, and the use of a computer based decision support system to facilitate the diagnosis and treatment of cancer related pain.

Primary hypothesis is, that this approach improves pain control and pain management in an unselected group of cancer patients in an outpatient setting.

* Improvement of average pain last 24 hours by at least 1.5 points on a 0-11 scale
* Improvement of worst pain last 24 hours by at least 1.5 points on a 0-11 scale
* An alteration in the prescribing dose of opioids in equipotent opioid dosage

Secondary hypothesis is, that this system improves overall symptom control and symptom management in an unselected group of cancer patients in an outpatient setting.

DETAILED DESCRIPTION:
The traditional way of symptom assessment is by the paper-and-pen method, which suffers from several limitations. The assessment items are not individually adjusted to each patient and his/her subjective symptoms, the collected data is rarely used in clinical practice, and decision-support for the physician is not possible.

Although the body of evidence is accumulating regarding the benefits of computerised symptom assessment in cancer patients, there is still insufficient knowledge of the impact of computerised assessment tools on the management of cancer pain and other cancer related symptoms.

The COMBAT study aims to investigate if a computer based assessment of cancer related symptoms, and a computerized decision support can improve treatment of pain and other symptoms in cancer patients.

This is an open, comparative study with a sequential design with two consecutive study periods, the non-intervention period and the intervention period.

The computer-based clinical decision support system will utilize the following data to generate one or several treatment options:

1. Data from self assessment of cancer related symptoms
2. Data from relevant variables reported by the physician
3. Revisited guidelines on treatment of cancer pain

ELIGIBILITY:
Inclusion Criteria:

* attending the outpatient clinic at the Cancer Clinic, St. Olavs Hospital Trondheim
* histologically verified malignancy
* able to follow study instructions
* able to read the information on the computer screen in the intervention period of the study
* able to use a touch screen in the intervention period of the study
* cancer related pain measured as average pain in last 24 hours of 4 or above on a numeric rating scale
* elective or emergency consultation with a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
average and worst pain during the last 24 hours | 1 week
  - The Brief Pain Inventory (BPI, a self-reported pain assessment tool aiming to quantify two aspects of cancer pain: Pain intensity and the functional disability as a result of cancer pain.
average and worst pain during the last 24 hours | 3 weeks
  - The Brief Pain Inventory (BPI, a self-reported pain assessment tool aiming to quantify two aspects of cancer pain: Pain intensity and the functional disability as a result of cancer pain.
average and worst pain during the last 24 hours | 1 week
  - The Alberta Breakthrough Pain Assessment Tool for cancer patients (ABPAT), a questionnaire developed in order to measure several dimensions of cancer-related breakthrough pain. It contains 15 questions, and was translated into Norwegian by our research group according to EORTC's rules for translation.
average and worst pain during the last 24 hours | 3 weeks
  - The Alberta Breakthrough Pain Assessment Tool for cancer patients (ABPAT), a questionnaire developed in order to measure several dimensions of cancer-related breakthrough pain. It contains 15 questions, and was translated into Norwegian by our research group according to EORTC's rules for translation.

SECONDARY OUTCOMES:
symptoms | 1 week
  - The Edmonton Symptom Assessment System (ESAS), a validated standardized questionnaire consisting of 10 items, which evaluate physical and psychological symptoms as well as general wellbeing.
symptoms | 3 weeks
  - The Edmonton Symptom Assessment System (ESAS), a validated standardized questionnaire consisting of 10 items, which evaluate physical and psychological symptoms as well as general wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Oncology outpatient clinic, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Raj SX, Brunelli C, Klepstad P, Kaasa S. COMBAT study - Computer based assessment and treatment - A clinical trial evaluating impact of a computerized clinical decision support tool on pain in cancer patients. Scand J Pain. 2017 Oct;17:99-106. doi: 10.1016/j.sjpain.2017.07.016. Epub 2017 Aug 8. PMID 28850380